CLINICAL TRIAL: NCT04537416
Title: Multidisciplinary Team-Based Study to Optimize the Evaluation and Treatment of Women With Thrombophilia and Recurrent Pregnancy Loss
Brief Title: Fertility, Hypercoagulability, and Inflammation (FREYA) Registry
Acronym: FREYA
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Associate Director, Thrombosis Research Group, Brigham and Women's Hospital
Other Study IDs: 2017P001215/PHS
Record Dates: First submitted 2020-08-29; First posted 2020-09-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Thrombophilia
MeSH Terms: conditions — Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with recurrent pregnancy loss: consecutive women at least 18 years old but not greater than 40 years old with a chief complaint of recurrent pregnancy loss
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A PubMed search of "thrombophilia" and "infertility" yields only 98 articles, the majority found in foreign medical journals and subspecialty journals with narrow readerships. Outside of Assisted Reproduction Clinics at academic medical centers, health care providers have limited awareness of the literature supporting thrombophilia evaluation and treatment in patients with recurrent pregnancy loss. As a result, women may suffer through years of repeated miscarriages before a thrombophilia evaluation is performed. By the time thrombophilia has been diagnosed as the cause of recurrent pregnancy loss, couples have often exhausted their personal savings on costly assisted reproductive therapies and present frustrated and psychologically exhausted.

In this study, we will evaluate the frequency of thrombophilia as a cause of recurrent pregnancy loss and provide insights into our patient care experience at BWH.

DETAILED DESCRIPTION:
Study Design:

Over a 2-year period, we will perform a retrospective observational cohort analysis of 1000 patients referred to the BWH Center for Infertility and Reproductive Surgery for evaluation of recurrent pregnancy loss. This cohort will include a retrospective analysis of 200 infertility patients referred to Dr. Piazza's Cardiovascular Medicine clinic for evaluation of thrombophilia.

We will also enroll prospectively for 18 months patients referred to the BWH Center for Infertility and Reproductive Surgery for evaluation of recurrent pregnancy loss.

Study Population:

We will include a study population that is representative of the ethnic and racial diversity of women who receive care at BWH. We will not enroll post-menopausal women, men or children because recurrent pregnancy loss specifically affects women of child-bearing potential. We do not plan to enroll pregnant women because we are specifically focused on women with recurrent pregnancy loss presenting for assisted reproductive therapy.

Retrospective Cohort:

For our retrospective analysis we will include 800 consecutive women at least 18 years old but not greater than 40 years old with a chief complaint of recurrent pregnancy loss referred to the BWH Center for Infertility and Reproductive Surgery and 200 consecutive patients referred to Dr. Piazza's Cardiovascular Medicine clinic for evaluation of thrombophilia as a cause of recurrent pregnancy loss. This will provide a total of 1000 patients for the retrospective cohort analysis.

Study Inclusion Criteria

1. Age 18-40 years
2. 2 or more pregnancy losses (including chemical pregnancies but not ectopic pregnancy)
3. Evaluated at the BWH Center for Infertility and Reproductive Surgery or the Watkins Cardiovascular Clinic

Study Exclusion Criteria

1. Infertility due to uterine factors (such as Asherman's Syndrome)
2. Known translocation carrier
3. Prior venous thromboembolism on anticoagulation
4. Abnormal uterine cavity on hysterosalpingogram/hysteroscopy

Prospective Cohort:

For the 18-month prospective cohort analysis, we will enroll consecutive patients evaluated at the BWH Center for Infertility and Reproductive Surgery for recurrent pregnancy loss.

Study Inclusion Criteria

1. Age 18-40 years
2. 2 or more pregnancy losses (including chemical pregnancies but not ectopic pregnancy)
3. Evaluated at the BWH Center for Infertility and Reproductive Surgery

Study Exclusion Criteria

1. Infertility due to uterine factors (such as Asherman's Syndrome)
2. Known translocation carrier
3. Prior venous thromboembolism on anticoagulation
4. Abnormal uterine cavity on hysterosalpingogram/hysteroscopy

Study Procedures:

From the EPIC Electronic Health Record (EHR), we will record demographic characteristics, comorbid conditions, details about the presentation of infertility, pregnancy losses, and prior assisted reproductive treatments, thrombophilia panel results, treatments, and outcomes, including successful pregnancies and deliveries. We will calculate the prevalence of thrombophilia in patients referred to BWH Center for Infertility and Reproductive Surgery for evaluation of recurrent pregnancy loss. We will describe the outcomes of patients receiving prophylactic low-dose anticoagulation, including bleeding, thrombotic events, and live births. We will perform multivariable regression analyses to answer additional key questions of predictors of thrombophilia as a cause of recurrent pregnancy loss and successful treatment of infertility due to thrombophilia.

The proposed retrospective and prospective cohort analysis will provide information about the standard of care at BWH for patients with recurrent pregnancy loss who may have thrombophilia. The registry will not change the standard of care for diagnosis and treatment of the patients at BWH in any way. The registry will not mandate any testing or treatments. There will be no required study visits, follow-up, or subject or provider contact.

Data Analysis Plan:

We will describe the results of patients receiving prophylactic anticoagulation, including frequency of bleeding and thrombotic events. We will calculate the prevalence of thrombophilia in patients referred to BWH Center for Infertility and Reproductive Surgery for evaluation of recurrent pregnancy loss. We will perform multivariable regression analyses to answer additional key questions of predictors of thrombophilia as a cause of recurrent pregnancy loss, chemical pregnancy after assisted reproductive therapy, and successful treatment of infertility due to thrombophilia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40 years
2. 2 or more pregnancy losses (including chemical pregnancies but not ectopic pregnancy)
3. Evaluated at the BWH Center for Infertility and Reproductive Surgery or the Watkins Cardiovascular Clinic

Exclusion Criteria:

1. Infertility due to uterine factors (such as Asherman's Syndrome)
2. Known translocation carrier
3. Prior venous thromboembolism on anticoagulation
4. Abnormal uterine cavity on hysterosalpingogram/hysteroscopy

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — It is a study on miscarriage. Hence can only be women.
Study Population: Women at least 18 years old but not greater than 40 years old with a chief complaint of recurrent pregnancy loss
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of laboratory diagnosed thrombophilia | 1 year
  Laboratory diagnosed acquired or inherited thrombophilia

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No